CLINICAL TRIAL: NCT02597101
Title: Neutrophil Elastase Inhibition as Adjunctive Therapy to Improve Glucometabolic Variables in Overweight and Obese, Insulin-Resistant Type 2 Diabetic Patients
Brief Title: Anti-Inflammatory Small Drug Adjunctive Therapy for Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nick Giannoukakis, PhD (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Pittsburgh (Other); University of South Florida (Other); AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Nick Giannoukakis, PhD, Associate Professor of Immunology and Biological Sciences, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Organization: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC-6059; 1UH3TR001372-01 (NIH)
Record Dates: First submitted 2015-11-03; First posted 2015-11-05 (Estimated); Results first posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Type 2 Diabetes Mellitus; Insulin Resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Metformin; saxagliptin; N-((5-(methanesulfonyl)pyridin-2-yl)methyl)-6-methyl-5-(1-methyl-1H-pyrazol-5-yl)-2-oxo-1-(3-(trifluoromethyl)phenyl)-1,2-dihydropyridine-3-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 5 mg saxagliptin, once a day, together with optimised (after titration) metformin (500-2000 mg/day) and 60 mg placebo tablet twice daily
  Interventions: Drug: Metformin; Drug: saxagliptin; Drug: placebo
- AZD9668 (Experimental): 60 mg AZD9668 twice daily in addition to 5 mg saxagliptin, once a day, together with optimised (after titration) metformin (500-2000 mg/day)
  Interventions: Drug: Metformin; Drug: saxagliptin; Drug: AZD9668

INTERVENTIONS:
Drug: Metformin — background drug
Drug: saxagliptin — background drug
  Other Names: onglyza
Drug: AZD9668 — study drug
  Arms: AZD9668
Drug: placebo — placebo for AZD9668 to be added to background drugs
  Arms: Placebo

SUMMARY:
The role of individual leukocyte populations in type 2 diabetes (T2D) and immunometabolism in general represent important gaps in knowledge to better understand the etiopathogenesis of T2D. Emerging evidence indicates that certain leukocyte populations serve as an important nexus of T2D-associated inflammation. This novel and innovative clinical trial will test the efficacy of a leukocyte-selective anti-inflammatory small drug as adjunctive therapy in improving insulin sensitivity in obese, insulin-resistant type 2 diabetic subjects. This trial also offers a first-in-kind opportunity to better understand the role of specific leukocyte populations in type 2 diabetes. The drug's clinical profile suggests that it will be well-tolerated with few, if any, side effects, and the existence of simple methods that can indirectly measure its activity in vivo

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) is characterized by concomitant insulin resistance and pancreatic beta cell dysfunction. Disease prevalence continues to increase around the globe and is currently estimated to be at more than 385 million affected people. As many as 1 in 3 people in the United States could have diabetes by the year 2050 with significant economic consequences. In 2014, 1 in 5 health care dollars was spent to support the care of patients at a total estimated cost > $245 billion. Overweight, insulin-resistant (IR) T2D individuals manifest a chronic systemic inflammation which impairs beta cells and peripheral insulin sensitivity. This systemic inflammation is associated with an atherogenic lipid profile and predisposes individuals to higher risk for micro- and macro-vascular disease, irrespective of well-controlled glycemia. Although a variety of pharmacologic approaches maintain daily glycemic control, it is becoming evident that there is an urgent need to identify adjunctive therapies to improve, insulin sensitivity, beta cell function, and HbA1c since they begin deteriorating quite substantially by 5 years following initial treatment. Ideally, such adjunctive therapies should be well-tolerated, easy to administer, should not promote hypoglycemia and should also attenuate the systemic inflammation. The role of neutrophils in T2D and metabolic inflammation represents an important gap in knowledge to better understand inflammation in T2D especially since neutrophils are the most abundant leukocyte population in humans and constitute the bulk of inflammatory leukocytes. Emerging evidence indicates that neutrophils along with neutrophil-derived elastase serve as an important nexus of T2D-associated inflammation. This trial offers a first-in-kind opportunity to better understand the role of neutrophils in T2D diabetics. We hypothesise that inhibition of neutrophil elastase (NE) will attenuate the chronic systemic background inflammation in overweight and obese, IR T2D subjects and that the potential improvement in insulin sensitivity and glucose control could concurrently facilitate functional maintenance and induce the rescue of pancreatic beta cell mass.

To test the hypothesis, we propose a clinical trial that is comprised of the following two aims:

Aim 1: To test whether orally-administered NEI adjunctive therapy in obese, IR T2D subjects improves insulin sensitivity, glucoregulation and glycemic control. The primary endpoint is the improvement of insulin sensitivity at 6 months compared to baseline, assessed by the hyperinsulinemic-euglycemic clamp method. Secondary endpoints will include: i) Safety (rate and severity of adverse events including hypoglycemia); ii) Glycemic and metabolic control variables; iii) Assessment of functional beta cell mass (improvement in baseline oral glucose tolerance test (OGTT) C-peptide levels and AUC, insulin secretion rate (ISR), body mass and body fat-corrected insulin sensitivity; and iv) Changes in inflammatory variables. Exploratory endpoints will include improvement of OGTT C-peptide (and C-peptide AUC) trajectory, ISR trajectory, and decreased dose and dose frequency of background drugs.

Aim 2: To inform the changes in innate and cellular immunity conferred by the trial study agents as a mechanistic approach to understanding the basis of potential efficacy. Evidence of suppression of systemic inflammation will be examined during the trial. Changes in gene expression of PBL and neutrophils may provide a signature of responder versus non-responder status and/or of effect of therapy.

ELIGIBILITY:
INCLUSION CRITERIA

1. Patients 21-75 years of age inclusive who meet the American Diabetes Association standard criteria for type 2 diabetes mellitus (T2D).
2. Subjects are currently on metformin (at least 1000 mg per day) for a minimum period of 4 weeks prior to screening visit alone, or in combination with any of the following diabetes medications or combinations:

   1. DPPIV inhibitor (any dose level/frequency)
   2. Sulfonylurea (any dose level/frequency)
   3. GLP1 agonist (any dose level/frequency)
   4. Sulfonylurea (any dose level/frequency) + GLP1 agonist (any dose level/frequency)
   5. Meglitinide (any dose level/frequency)
   6. SGLT2 inhibitor (any dose level/frequency)
3. Patients must have a body-to-mass index (BMI) of greater than or equal to 27 kg/m2.
4. Patients exhibit glycated HbA1c between 7.3-11.0 during eligibility screening and then <=8.5 at final run-in visit.
5. Willingness to replace current diabetes therapies (listed in inclusion 2) with metformin and saxagliptin and to adjust metformin dose during run-in period.
6. Subjects present adequate immune competence as assessed by immunoreactivity to viral antigens (CEF Pool Assay) in vitro at the time of screening.
7. Participants of childbearing potential must agree to practice an effective form of birth control which may include any one of the following: barrier method, oral contraception, or surgery. These measures must be maintained throughout the study.
8. Subjects must have good peripheral venous access for the hyperinsulinemic-euglycemic clamp and the 3-hr. OGTT procedures.
9. Patients understand the study procedures, alternative treatments available, risks involved in the study, and voluntarily agree to participate by giving informed and signed written consent for screening and enrollment.
10. Participants can be on anti-inflammatory therapies that are not diabetes-focused (e.g. non-salicylate anti-inflammatory therapies, non-salicylate NSAIDs) and/or anti-hypertensive medicaments or statins.

EXCLUSION CRITERIA

1. Patients with type 1 diabetes mellitus as defined by the American Diabetes Association criteria or a history of ketoacidosis, or the patients are assessed by the study team as possibly having type 1 diabetes mellitus confirmed with the presence of at least one of the typical autoantibodies (insulin, GAD65, IA-2, ZnT8) AND a serum C-peptide level of <0.7 ng/mL.
2. Patients have been treated with any therapies specific for their diabetes (other than those listed in the inclusion criteria) within 4 weeks of the screening visit.
3. Patients have been treated with insulin within 2 months of the screening visit.
4. Patients are currently participating in or have participated in another study with an investigational compound or device within the prior 12 weeks of signing the informed consent or do not agree to refrain from participating in any other study while participating in this study.
5. Patients have a history of hypersensitivity or any contraindication to DPPIV inhibitors, including saxagliptin (Onglyza), or metformin based upon the labels of the USA.
6. Patients are on a weight loss medication (such as orlistat, phentermine, Qsymia, or Belviq) within the prior 6 weeks.
7. Patients are required by treating physicians to remain on any one of these agents during the trial:

   macrolide antibiotics, cisapride, anti-arrhythmics, steroids, rifampicin, phenobarbital, phenytoin, secobarbital, carbamazepine, norethindrone, isoniazid. AZD9668 is metabolized by CYP3A4, 3A5, and 2B6. SAXA is metabolized by CYP3A4 and 3A5, potentially leading to drug-drug interactions with hypothetical adverse events in patients on the above agents. Also, AZD9668 causes weak inhibition of CYP2C9 and therefore patients on fluconazole, amiodarone, fenofibrate, fluvoxamine, phenylbutazone, probenecid, sertraline, will also be excluded to avoid the hypothetical adverse events due to this effect.
8. Patients have undergone major surgery within the 6 weeks prior to signing consent or have any type or form of major surgery planned during the study (at the discretion of the physician).
9. Patients are on or are likely to require treatment with 14 consecutive days or repeated courses of pharmacologic doses of corticosteroids or any other immunomodulatory agent. For example, patients requiring chronic systemic corticosteroids (does not include topical or inhaled corticosteroids). Exceptions are over the counter non-salicylate NSAIDs.
10. Enrollment or history of enrollment in a drug, or biologic therapy clinical trial that affects the immune system within the past 12 months (e.g., systemic immunosuppressive pharmacologics, immunosuppressive cytokines, therapeutic immunomodulating antibodies, therapeutic immunomodulating fusion proteins and/or cytokine receptor decoys as well as any intervention and/or non-intervention induced immunodeficiencies).
11. Prior history of coronary artery disease (defined as myocardial infarction, angina, bypass surgery, or angioplasty)
12. Prior history of arrhythmia (excludes premature beats)
13. Prior history of heart failure defined as i) symptomatic OR ii) pulmonary edema, leg edema or low ejection fraction (<40%)
14. Evidence of refractory chronic migraine (defined in ICHD-3 and Martelletti et al.).
15. History of persistent bradycardia within the last year prior screening visit (more than three episodes in a calendar year of a heart rate <60 beats per minute that required hospitalization on each of these occasions).
16. Leukopenia (<3000 leukocytes/microliter), neutropenia (1500 neutrophils/microliter), lymphopenia (<800 lymphocytes/microliter), or thrombocytopenia (<125000 platelets/microliter),. any other clinically relevant abnormal hematology value.
17. Positivity for HIV, active CMV, chlamydia, any evidence of serious fungal infection, active HSV1and/or HSV2 (determined as IgM positivity of 2 standard deviations higher than the highest value of the test reference range), hepatitis B or C, at screening. Minor skin fungus, or minor candidiasis is not an enrollment or treatment exclusion criterion. Also, with the exception of HIV history, hepatitis B and C, successfully-treated, disease-free individuals (> 6 months between time of successful treatment confirmation and time at screening) would be eligible for enrollment in this trial.
18. Patients are required by treating physician to remain on any medications listed in inclusion #2 that directly affect glucose metabolism such as, but not limited to thiazolidinediones, pramlintide, or amylin.
19. Vaccination with any form of live vaccine product within the last 3 months prior to initiation of study agent administration.
20. Any chronic disease that in the opinion of the investigators would affect the patient's safety and/or the integrity of the study outcome. This does not include dyslipidemia, patients on statin or anti- hypertension treatment, or patients with well-controlled hypo- or hyperthyroidism
21. Any other disease or disorder requiring chronic drug therapy except for treated hypothyroidism (T4 and TSH should be within the normal reference range adjusted for age), celiac disease, or statin- maintained, uncomplicated lipidemia.
22. Evidence of liver dysfunction, with ALT or AST> 1.5 times the upper limit of normal.
23. Evidence of renal insufficiency as indicated by blood creatinine of > 2 times the upper limit of normal at baseline screening OR an eGFR < 45 mL/min. OR A past history or current clinical evidence of renal failure or low creatinine clearance at screening.
24. Females who are pregnant at the time of screening or unwilling to defer pregnancy during the study period.
25. Lactating women.
26. Poor accessibility to veins for the 3-hour OGTT and hyperinsulinemic-euglycemic clamp procedures.
27. The following therapies cannot be administered while patients are undergoing treatment on this protocol: i) radiation therapy; ii) chemotherapy; iii) corticosteroids (except for very short courses of topical or inhaled); iv) agents used to treat attention deficit and hyperactivity disorder (ADHD); v) rifampicin or phenytoin; vi) other protein, particle or cell vaccine immunomodulation therapies. If these therapies are essential for treatment of other conditions, participation in this study will be terminated.
28. A condition which interferes with the ability to accurately determine glycated HbA1c. Examples include: Genetic variants (e.g. HbS trait, HbC trait), elevated fetal hemoglobin (HbF) and chemically modified derivatives of hemoglobin (e.g. carbamylated Hb in patients with renal failure); Any condition that shortens erythrocyte survival or decreases mean erythrocyte age (e.g., recovery from acute blood loss, hemolytic anemia); Iron deficiency anemia, iron replacement therapy
29. Subjects who cannot tolerate at least 1000 mg daily of immediate or extended release metformin by the time of final run-in will be excluded from further participation.
30. Subjects who do not exhibit a glycated HbA1c level <=8.5 by the end of the run-in period.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-11; Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nick Giannoukakis, Ph.D., Principal Investigator — Allegheny Health Network
Locations (1):
- Allegheny Health Network, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
While de-identified data (outcomes, measurements) from single study participants will be recorded and available through requests to the NIH, publicly-available data will be in the form of means, medians, and descriptive aggregate values representing the treatment groups in peer-reviewed publications.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Immediate (as of January 29, 2021); available until January 31, 2031.
Access Criteria: Upon request to the Study PI.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 14 subjects consented (9 screen failures, 5 randomized). Of the 5 randomized, 4 completed both arms while 1 was withdrawn after completing the AZD9668 arm and did not crossover to placebo.
Period: Overall Study
Arm/Group | Placebo | AZD9668
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | AZD9668 | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 9
Insulin Sensitivity [Mean (Standard Deviation); unit: (ml/kg/min)/(microIU/ml)] — Insulin sensitivity at baseline, assessed by the hyperinsulinemic-euglycemic clamp method.
  M/LBM = whole-body insulin sensitivity adjusted for lean body mass. M/LBM is calculated as the steady-state glucose disposal (in mL) per kilogram lean body mass divided by steady-state insulin concentrations (micro IU/mL).
  (ml/kg/min)/(microIU/ml) | 8.05 (7.4) | 9.9 (3.3) | 8.975 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity at 6 Months From Baseline
Description: The primary outcome measure is the insulin sensitivity at 6 months from baseline, assessed by the hyperinsulinemic-euglycemic clamp method. This is calculated as the M/LBM. M/LBM = whole-body insulin sensitivity adjusted for lean body mass. M/LBM is calculated as the steady-state glucose disposal (in mL) per kilogram lean body mass divided by steady-state insulin concentrations (micro IU/mL).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: (mL/kg/min)/(microIU/mL)
Arm/Group | Placebo | AZD9668
Number analyzed (Participants) | 4 | 5
(mL/kg/min)/(microIU/mL) | 9.9 (3.7) | 6.4 (3.5)
Statistical Analysis 1: Comparison: Placebo vs AZD9668; The primary efficacy endpoint is the improvement of insulin sensitivity by 40% or greater at 6 months compared to baseline, assessed by the hyperinsulinemic-euglycemic clamp method; Test type: Other — REML mixed model; p < 0.05, REML mixed model — Using REML mixed model analysis, differences between study arms resulting in a p<0.05 would represent statistically-significant differences; REML mixed model = 0.05

2. Secondary Outcome: Severity of All Adverse Events Including Hypoglycemia
Description: Severity of all adverse events including hypoglycemia based on the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 severity grade score (0-4). Higher scores indicate a worse severity.
Time Frame: 12 months
Population: Full Analysis Set
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AZD9668
Number analyzed (Participants) | 4 | 5
score on a scale | 0 (0) | 0 (0)

3. Secondary Outcome: Severity of Known AEs of AZD9668
Description: Attribution score of AE to known AEs of AZD9668 in terms of an atribution scale of 0-4. The scale is defined as: Score 0=Unrelated; Score 1=The AE is unlikely related; Score 2=The AE has a reasonable possibility to be related; Score 3=The AE is likely related; Score 4=The AE is clearly related
Time Frame: 12 months
Population: Full Analysis Set
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AZD9668
Number analyzed (Participants) | 4 | 5
score on a scale | 0 (0) | 0 (0)

4. Secondary Outcome: Severity of Known AEs of Saxagliptin
Description: Attribution score of AE to known AEs of saxagliptin in terms of an atribution scale of 0-4. The scale is defined as: Score 0=Unrelated; Score 1=The AE is unlikely related; Score 2=The AE has a reasonable possibility to be related; Score 3=The AE is likely related; Score 4=The AE is clearly related
Time Frame: 12 months
Population: Full Analysis Set
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AZD9668
Number analyzed (Participants) | 4 | 5
score on a scale | 0 (0) | 0 (0)

5. Secondary Outcome: Severity of Known AEs of Metformin
Description: Attribution score of AE to known AEs of metformin in terms of an atribution scale of 0-4. The scale is defined as: Score 0=Unrelated; Score 1=The AE is unlikely related; Score 2=The AE has a reasonable possibility to be related; Score 3=The AE is likely related; Score 4=The AE is clearly related
Time Frame: 12 months
Population: Full Analysis Set
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AZD9668
Number analyzed (Participants) | 4 | 5
score on a scale | 0 (0) | 0 (0)

6. Secondary Outcome: Change in Glycated HbA1c Levels Compared to Baseline
Description: Difference in the value of HbA1c study end (12 months) compared to baseline value (time 0)
Time Frame: 12 months
Population: ITT
Measure: Mean (Standard Deviation); unit: percentage of the change from baseline
Arm/Group | Placebo | AZD9668
Number analyzed (Participants) | 4 | 5
percentage of the change from baseline | 7.2 (1.4) | 7.6 (0.9)

7. Secondary Outcome: Change in OGTT From Baseline
Description: The difference of the calculated area under the curve of the 2 hour OGTT test (AUC is the value of the area under the glucose concentration time curve) at 12 months minus the AUC at baseline (time zero). This AUC is calculated as the concentration of glucose versus time curve and the reporting units are mcg*dL/hour. The trapezoid rule was applied to the curve to obtain the AUC.
Time Frame: 12 months
Population: ITT
Measure: Mean (Standard Deviation); unit: mcg*dL/hour
Arm/Group | Placebo | AZD9668
Number analyzed (Participants) | 4 | 5
mcg*dL/hour | 732.9 (156.6) | 821.4 (185.2)

8. Secondary Outcome: Change in OGTT-derived Insulinogenic Index Using C-peptide
Description: The change from baseline at 12 months where the insulinogenic index = ratio of fasting C-peptide concentration (ng/mL)/fasting glucose (ng/mL) at the time of the OGTT test.
Time Frame: 12 months
Population: ITT
Measure: Mean (Standard Deviation); unit: ratio of fasting C-peptide concentration
Arm/Group | Placebo | AZD9668
Number analyzed (Participants) | 4 | 5
ratio of fasting C-peptide concentration | 21.9 (2.2) | 22.6 (5.2)

9. Secondary Outcome: Change From Baseline in the Serum Levels of Inflammatory Markers
Description: Serum levels refers to the concentration in serum of each of the analytes in the multi-analyte assay (Luminex) in terms of pg/mL depending on the analyte measured. We are reporting the difference in these values between 12 months and baseline.
Time Frame: 12 months
Population: ITT
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | AZD9668
Number analyzed (Participants) | 4 | 5
pg/mL
  Eoatxin | 33.1 (20.9) | 39.2 (23.2)
  GM-CSF | 8.8 (0.3) | 8.8 (0.3)
  INFa | 17.6 (4.6) | 18.8 (4.6)
  IL-1RA | 75.3 (14.6) | 87.6 (34.0)
  IL-2 | 5.3 (0.1) | 5.3 (0.2)
  IL-2R | 208.6 (94.9) | 167.1 (107.1)
  IL-4 | 22.6 (1.1) | 22.4 (1.1)
  IL-5 | 4.8 (1.1) | 4.7 (0.9)
  IL-6 | 3.4 (0.7) | 3.2 (0.4)
  IL-7 | 10.4 (8.2) | 9.0 (6.4)
  IL-8 | 8.0 (2.0) | 8.2 (0.7)
  IL-10 | 11.2 (0.4) | 11.3 (0.6)
  IL-12 | 44.3 (12.1) | 43.4 (22.7)
  IL-13 | 12.0 (1.8) | 12.0 (1.8)
  IL-15 | 50.9 (14.4) | 47.7 (18.5)
  IL-17 | 11.0 (0.8) | 10.8 (0.6)
  INFy | 20.1 (4.7) | 17.8 (5.8)
  IP-10 | 25.2 (17.2) | 19.7 (17.5)
  MCP-1 | 71.0 (29.5) | 93.5 (25.2)
  MIG | 13.9 (9.4) | 22.1 (22.2)
  MIP-1a | 14.8 (2.2) | 14.6 (2.9)
  MIP-1b | 69.1 (27.9) | 81.5 (30.3)
  RANTES | 532.6 (612.5) | 219.5 (125.9)
  TNFa | 10.9 (3.3) | 10.7 (3.3)

ADVERSE EVENTS:
Time Frame: 12 months
Description: The definition of AE/SAE used to collect AE information does not differ from the clinicaltrials.gov definitions.
Arm/Group | Placebo | AZD9668
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5

LIMITATIONS AND CAVEATS:
The failure to enroll a critical mass of study subjects renders the outcome difficult to interpret given the inability to conduct statistical analyses that would be more meaningful.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-06-13): https://cdn.clinicaltrials.gov/large-docs/01/NCT02597101/Prot_SAP_ICF_000.pdf